CLINICAL TRIAL: NCT02336646
Title: Cell Therapy With Mesenchymal Stem Cell in Ischemic Limb Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Bio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-02-070B
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2015-11

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Allogenic MSC (Experimental): Low dose allogenic mesenchymal stem cells with IM injection
  Interventions: Drug: Allogenic MSC
- High Dose Allogenic MSC (Experimental): High dose allogenic mesenchymal stem cells with IM injection
  Interventions: Drug: Allogenic MSC
- Placebo (Placebo Comparator): normal saline with Intramuscular injection
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Allogenic MSC — Hypoxia-cultured human bone marrow derived mesenchymal stem cells
  Other Names: Biochymal
  Arms: High Dose Allogenic MSC; Low Dose Allogenic MSC
Drug: Normal saline
  Arms: Placebo

SUMMARY:
Bone marrow MSCs will be isolated from allogenic donors, expanded under hypoxic conditions using medium containing no serum or animal-derived reagents, and applies for Phase Ⅰ/Ⅱ study in treating 18 recipients with ischemic limb diseases.

DETAILED DESCRIPTION:
Ischemic limb disease remains one of the major causes of morbidity and mortality in the industrialized world despite the development of several new therapeutic modalities. Based on experimental data demonstrating that infusion or injection of stem/progenitor cells enhances blood flow in models of cardiovascular diseases, clinical trials were initiated in 2001 to treat patients with critical limb ischemia or cardiac ischemia with circulating blood or bone marrow-derived cells. Despite all promises, pending uncertainties and practical limitations attenuate the therapeutic use of stem/progenitor cells for ischemic limb disease. The main theme and method in the current program project, based on expertise, track record, and preliminary results of PI's laboratory, is to focus on clinical studies of using allogenic mesenchymal stem cells (MSCs), expanded under hypoxic conditions (1% O2), in treating ischemic limbs. This project is an integrated and coordinated effort aimed to overcome the regulation of cell product, and the barriers of preclinical and clinical studies. For the purposes, we have specially set up the core laboratory for stem/progenitor cells production and quality control in Cell Therapy Clean Room on the 9th floor of Medical Science Technology Building in Taipei Veterans General Hospital. We have also completed the preclinical studies in using allogenic hypoxic mouse MSCs in treating limb ischemia. In the current project, bone marrow MSCs will be isolated from allogenic donors, expanded under hypoxic conditions using medium containing no serum or animal-derived reagents, and applies for Phase Ⅰ/Ⅱ study in treating 18 recipients with ischemic limb diseases in three years.

ELIGIBILITY:
Inclusion Criteria:

* Fontaine stage > II, total walking distance < 100 m, stair < 1 floor, or ulcer / necrosis
* Established critical limb ischemia, clinically and hemodynamically confirmed as per Rutherford- Ⅱ-4, Ⅲ-5, or Ⅲ-6; Patients having Infra-inguinal arterial occlusive disease with rest pain or ischemic ulcer/necrosis, who are not eligible for or have failed traditional revascularization treatment
* Ankle Brachial Pressure Index (ABPI) ≤ 0.8，ankle pressure ≤ 70 mm Hg, or TcPO2 ≤ 70 mmHg in the foot
* No response to medication (aspirin and cilostazol)
* Normal liver and renal function
* On regular medication for hypertension if any

Exclusion Criteria:

* The above mentioned patients combined with infection or systemic septicemia. (ps, patients with poor control of diabetes, hypertension and hyperlipidemia will also be excluded
* Patient with Immunocompromised or immunosuppressed
* Type I Diabetes
* Patients having stroke or myocardial infarction within last 3 months
* Hb% < 10 gm%, Serum Creatinine ≥ 2mg%, Serum Total Bilirubin ≥2mg%, HbA1c > 8%

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months
  Number of adverse events reported

SECONDARY OUTCOMES:
Efficacy-The Wong Baker FACES® pain rating scale | 6 months
  The Wong Baker FACES® pain rating scale, for evaluation of ischemic pain in the diseased lower limb of subjects receiving cell injection compared to placebo
Efficacy-Transcutaneous oxygen pressure(TcPO2) | 6 months
  The Transcutaneous oxygen pressure (TcPO2) on foot of subjects receiving cell injection compared to placebo
Efficacy-walking distance (TWD) | 6 months
  Total walking distance (TWD) on a standardized treadmill test compared to placebo
Efficacy-Ankle Brachial Pressure Index (ABPI) | 6 months
  The Ankle Brachial Pressure Index (ABPI) in the lower limb of subjects receiving cell injection compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Chun Che Shih, Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan